CLINICAL TRIAL: NCT03191851
Title: Evaluation of 'Melody' Paracentesis Device for Ascites Therapy in Patients With Cirrhosis (EMPATHY)
Brief Title: Evaluation of 'Melody' Paracentesis Device for Ascites Therapy
Acronym: EMPATHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Mediplus Ltd UK (Unknown); Enteric healthcare technology Co-operative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14083
Record Dates: First submitted 2016-12-01; First posted 2017-06-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Ascites Hepatic; Cirrhosis and Chronic Liver Disease
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Device (Active Comparator): Standard device
  Interventions: Device: standard device
- Melody Device (Experimental): Melody device without Pump
  Interventions: Device: Melody Device
- Melody Device with pump (Experimental): Melody Catheter device with Andromeda Pump
  Interventions: Device: Melody Device with Pump

INTERVENTIONS:
Device: standard device — paracentesis using standard
  Arms: Standard Device
Device: Melody Device — paracentesis using Melody Device
  Other Names: Melody Catheter
  Arms: Melody Device
Device: Melody Device with Pump — paracentesis using Melody Device with Pump
  Other Names: Melody Catheter with Andromeda Pump
  Arms: Melody Device with pump

SUMMARY:
Ascites is the accumulation of fluid inside the abdomen. This can happen when the liver fails due to a substantial amount of scarring (cirrhosis). Patients (pts) must have this fluid drained and as cirrhosis progresses, patients will require drainage of ascites repeatedly on a regular basis, leading to frequent hospitals visits and increased complications.

The current drainage device is slow and doesn't always drain completely so pts have to return repeatedly to keep symptoms under control.

A new device (called Melody) has been developed and specifically designed for the purpose of draining ascites fluid, which the Investigators expect to drain faster and completely.

This study will compare the volume of ascites drained using the new 'Melody' catheter device with that used in standard NHS practice. If the melody catheter device is confirmed as superior to the current device this would improve patient experience (less frequent visits to hospital and increased length of time between visits).

With fewer procedures performed per patient, the pressure on the NHS would be greatly reduced in terms of time and costs.

DETAILED DESCRIPTION:
Large volume paracentesis has been established as a treatment for symptomatic ascites and is performed regularly in secondary care hospitals widely across the UK.

Lack of a device specifically designed to perform paracentesis means that flow of ascites fluid through the catheter is not optimal leading to incomplete drainage and hence, frequent repeated paracentesis as well as a number of complications.

A new 'Melody' catheter device has been designed and developed in collaboration with Mediplus Ltd and NIHR Enteric Bowel function Healthcare Technology Co-operative; specifically designed to improve the performance characteristics of paracentesis procedure.

(The 'Melody ascites drainage catheter' including 'sterile ascetic drainage sets' is CE marked for clinical use). In addition, investigators would also like to confirm whether the addition of a pump will improve drainage with this device further.

The Investigators propose to carry out a feasibility study, 'EMPATHY', with an aim to compare the performance characteristics of 'Melody' catheter device (with and without addition of 'Andromeda' pump) with the current device. 112 patients with ascites requiring therapeutic paracentesis will be randomised to undergo the procedure using one of the two devices. The volume of ascites drained per session will be compared along with ease of insertion and removal as well as patient experience including all adverse events up to 7 days following the procedure. The outcomes of this feasibility study will inform further refinement of the 'Melody' catheter device as well as a future large multi-centre randomised controlled trial evaluating the cost-effectiveness of the new 'Melody' catheter device in therapeutic paracentesis

ELIGIBILITY:
Inclusion Criteria:

* Ascites due to cirrhosis of the liver.
* Aged 18-80 years.
* Ability to give written consent.

Exclusion Criteria:

* Known untreated spontaneous bacterial peritonitis.
* Disseminated intravascular coagulation at the time of consenting.
* Pregnancy.
* Patients who have had more than six ascitic drainage procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Amount of ascites fluid drained (litres) | Up to 6 hours
  Amount of ascites fluid drained in one session (litres)

SECONDARY OUTCOMES:
Adverse Events | Up to 7 days
  As reported by patients using a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Guruprasad Aithal, Principal Investigator — NIHR Nottingham Biomedical Research Centre, Nottingham University Hospitals NHS Trust & University of Nottingham
Locations (1):
- Queen Day Case Unit Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No